CLINICAL TRIAL: NCT05316272
Title: Effects of DHEA and Exercise on Bone Marrow Fat in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 162427a; 5R01AR077924-03 (NIH)
Record Dates: First submitted 2022-03-17; First posted 2022-04-07 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Low Bone Density; Osteoporosis
MeSH Terms: conditions — Bone Diseases, Metabolic; Osteoporosis | interventions — Exercise; Dehydroepiandrosterone

STUDY DESIGN:
Intervention Model Description: Two-by-two crossed design of DHEA versus control and exercise versus no exercise control.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking of the study pill (DHEA or placebo) is described as noted above. Exercise cannot be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise and placebo (Experimental): supervised bone-loading exercise 3 days per week and one placebo pill per day for 36 weeks
  Interventions: Behavioral: Exercise; Dietary Supplement: DHEA
- Exercise and DHEA (Experimental): supervised bone-loading exercise 3 days per week and one dose of DHEA (50 milligrams) per day for 36 weeks
  Interventions: Behavioral: Exercise; Dietary Supplement: DHEA
- no exercise and DHEA (Experimental): no supervised bone exercise and one dose of DHEA (50 milligrams) per day for 36 weeks
  Interventions: Behavioral: Exercise; Dietary Supplement: DHEA
- no exercise and placebo (Experimental): no supervised bone-loading exercise and one placebo pill per day for 36 weeks
  Interventions: Behavioral: Exercise; Dietary Supplement: DHEA

INTERVENTIONS:
Behavioral: Exercise — Supervised bone-loading exercise on 3 days per week for 36 weeks
Dietary Supplement: DHEA — DHEA in pill form 50 milligrams taken daily for 36 weeks

SUMMARY:
Bone strength -the main determinant of bone fracture- is a function not only of bone mineral density (BMD) and microstructure, but also of its microenvironment, including bone marrow fat (BMF). The adrenal steroid dehydroepiandrosterone (DHEA) -the main precursor for estrogens and androgens in postmenopausal women- as well as bone-loading exercise, increase BMD in older women, however, their effects on BMF are largely unknown. This study has high potential to unveil the hormonal and mechanical effects of DHEA and exercise on BMF, respectively, and to elucidate longitudinal associations of BMF with bone strength in older women with bone loss.

DETAILED DESCRIPTION:
The proportion of the U.S. population older than 65 years will increase from 12.7% in 2000 to 20.3% in 2050, and the number of fractures is expected to exceed 3 million by 2025 with associated costs in the order of $25.3 billion per year. DAMES is an ongoing clinical trial (NCT03227458) that aims to assess -for the first time- changes in areal bone mineral density (aBMD) and fat-free mass (FFM) in response to therapy with the adrenal steroid dehydroepiandrosterone (DHEA) alone and combined with bone-loading exercise (EX) in older women with bone loss. The hormonal and mechanical strategies proposed in DAMES represent a low-cost alternative treatment to improve bone quantity with a number of other health benefits not afforded by typical pharmacological approaches. However, bone strength -the main determinant of bone fracture- is a function of not only BMD and microstructure, but also of its microenvironment, including bone marrow fat (BMF). This in an ancillary study to the DAMES clinical trial. Here, the investigators propose to leverage the well-characterized cohort of subjects, exercise training, clinical, laboratory and imaging data from DAMES, and add a small group of controls to its three existing arms (DHEA only, EX+Placebo, and EX+DHEA) to investigate the effects of DHEA therapy and EX on BMF in older women using advanced imaging, numerical engineering, and image analysis techniques. In particular, the investigators aim to determine in the lumbar spine and hip of older women with low bone mass or moderate osteoporosis: 1) whether DHEA or EX leads to changes in BMF content; 2) whether BMF content is associated with bone strength at baseline, and whether changes in BMF content are associated with changes in bone strength, evaluating the impact of DHEA or EX on these associations; and 3) the spatial distribution of changes in BMF content in response to DHEA or EX. BMF will be measured with chemical shift-based water-fat separation magnetic resonance imaging, bone strength will be estimated with finite element modeling from quantitative computed tomography scans, and differences in the spatial distribution of BMF changes between groups will be assessed using voxel-based morphometry. Ultimately, the investigators will leverage the DAMES clinical trial to unveil new information to improve our understanding of DHEA and EX on bone quantity and quality. The longitudinal assessments of bone quality in this ancillary proposal, with those of bone quantity in the parent study, in women who have already lost bone mass is unprecedented. Understanding how osteoporosis treatments -including exercise- act on BMF could lead to the generation of novel approaches for fracture risk assessment, procedures for therapy monitoring, and treatments for bone loss.

ELIGIBILITY:
Inclusion Criteria:

* women aged 55 to 85 years
* non-frail, as determined by Short Physical Performance Battery score > 9 (0-12 scale)
* 5 years or longer since menopause (defined as last menstrual period)
* willing to participate in a 36-week exercise program that will start at a moderate intensity and gradually progress to a higher intensity
* willing to take DHEA (50mg/d) or a placebo pill daily and remain blinded for up to 36 weeks
* not performing resistance exercise training or high impact weight-bearing exercise (e.g., jogging) ≥ 2 days per week in the past 6 months
* ambulatory without assistive devices
* serum DHEAS < 140 μg/dL (3.8 μmol/L)
* low bone mass or moderate osteoporosis indicated by lumbar spine, total hip, or femoral neck aBMD t-scores < -1.0 and ≥ -3.0
* refusal of standard osteoporosis treatment in women with moderate osteoporosis (BMD ≥-3.0 and ≤ -2.5)
* evidence of a negative (no findings suspicious for breast cancer) mammogram within the past 12 months
* planning to reside in the Denver area for the duration of the study
* willing to provide evidence of completed COVID-19 vaccination
* no implanted metal or electronic devices
* no metallic foreign body in the eye
* no "triggerfish" contact lenses
* no gastric reflux device
* no insulin pumps
* no temporary transvenous pacing leads
* no aneurysm clips
* no cardiac pacemakers
* no implanted cardioverter defibrillator
* no magnetically-activated implant or device
* no neurostimulation system
* no spinal cord stimulator
* no cochlear implant
* no bone growth/bone fusion stimulator
* no known claustrophobia

Exclusion Criteria:

* history of hospitalization for Corona Virus Disease 2019 (COVID-19)
* does not meet Centers for Disease Control and Prevention (CDC) recommendations for home isolation because has had a positive severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) test less than 10 days before study entry; or has had fever within the past 3 days and respiratory symptoms have not improved; or symptoms first appeared less than 10 days before study entry.
* not willing to provide evidence of completed COVID-19 vaccination.
* uncontrolled hypertension defined as resting systolic BP >150 mmHg or diastolic BP >90 mmHg; participants who do not meet these criteria at first screening will be re-evaluated, including follow-up evaluation by their primary care provider (PCP) with initiation or adjustment of anti-hypertensive medications.
* diagnosed ischemic heart disease or indicators of unstable ischemic heart disease (e.g., angina) or arrhythmias at rest or during the graded exercise test (GXT) without negative follow-up evaluation will be cause for exclusion; follow-up evaluation must include diagnostic testing (e.g., thallium stress test) with interpretation by a cardiologist
* diagnosis of heart failure, clinically significant aortic stenosis, uncontrolled angina, or uncontrolled arrhythmia.
* pulmonary disease requiring use of oral steroids within the previous 6 months or the use of supplemental oxygen ≥ 4 liters with physical exertion
* orthopedic problems (e.g., severe osteoarthritis, rheumatoid arthritis) that greatly limit the ability to perform moderate to high intensity resistance exercise (e.g., unable to be properly positioned in exercise equipment or to have severely restricted range of motion even after modifications have been made)
* hip fracture, hip or knee replacement, or spinal surgery in the past 6 months
* undergoing physical therapy involving the lower extremities
* hematocrit > 54%
* thyroid dysfunction, defined as an ultrasensitive thyroid stimulating hormone (TSH) < 0.4 or > 10 micro units/mL, without signs or symptoms of clinical hypo- or hyperthyroidism.volunteers with abnormal TSH values will be re-considered for participation in the study after follow-up evaluation by their PCP with initiation or adjustment of thyroid hormone replacement
* acute liver disease indicated by liver function tests (ALT, aspartate aminotransferase, alkaline phosphatase) ≥ 1.5 times the upper limits of normal
* estimated glomerular filtration rate (eGFR) < 45, using Modification of Diet in Renal Disease Study (MDRD) equation
* poorly controlled diabetes mellitus based on HbA1c > 8.5% or use of insulin.
* fasted serum triglycerides > 400 mg/dL
* serum 25-hydroxy vitamin D < 20 ng/mL; volunteers will be re-considered for participation in the study after initiation or adjustment of vitamin D supplementation, per the study's vitamin D repletion protocol.
* use of DHEA supplementation or sex hormones in the past 6 months. Use of prescription low dose vaginal estrogen creams (Premarin or Estrace) 3 days per week or less will not be exclusionary.
* use in the past 6 months of any medications known to alter bone metabolism (e.g., oral glucocorticoids, bone anti- resorptive agents)
* lumbar spine, total hip, or femoral neck aBMD t-scores < -3.0.
* confirmed history of osteoporotic fracture
* secondary osteoporosis
* documented history of cognitive impairment or dementia or Mini-Cog < 4.
* current smoker
* personal history of breast, ovarian, metastatic endometrial, or cervical cancer
* any cancer requiring treatment in the past 3 years except non-melanoma skin cancers
* undiagnosed vaginal bleeding
* women who, in the judgment of the study physician, appear incapable of safely participating in the exercise (e.g., neuromuscular/musculoskeletal impairment).
* Known claustrophobia if participating in the optional MRI study
* No metal implants (detailed above) if participating in the optional MRI study

Ages: 55 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in spine bone marrow fat content | 36 weeks
  changes in bone marrow fat content of the lumbar spine
Changes in hip bone marrow fat content | 36 weeks
  changes in bone marrow fat content of the proximal femur
Correlation of lumbar spine bone marrow fat content with bone strength at baseline | baseline - 0 weeks of intervention
  Correlation of lumbar bone marrow fat content (%) with strength (N) of the lumbar spine at baseline
Correlation of hip bone marrow fat content with hip strength at baseline | baseline - 0 weeks of intervention
  Correlation of proximal femur spine bone marrow fat content (%) with strength (N) of the proximal femur at baseline
Correlation of the changes in spine bone marrow fat content with changes in spine bone strength | 36 weeks
  Correlation of the changes in lumbar spine bone marrow fat content (%) with changes in lumbar spine strength (N)
Correlation of the changes in hip bone marrow fat content (%) with changes in hip bone strength (N) | 36 weeks
  Correlation of the changes in proximal femur bone marrow fat content (%) with changes in proximal femur bone strength (N)

OTHER OUTCOMES:
spatial distribution of the changes in bone marrow fat content of the spine | 36 weeks
  spatial distribution of the changes in bone marrow fat content of the lumbar spine
spatial distribution of the changes in bone marrow fat content of the hip | 36 weeks
  spatial distribution of the changes in bone marrow fat content of the proximal femur

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Jankowski, PhD, Principal Investigator — University of Colorado, Denver; Julio Carballido-Gamio, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No